CLINICAL TRIAL: NCT02182765
Title: An Investigation of the Potential Pharmacokinetic Interaction Between Nevirapine (VIRAMUNE®), Abacavir and Amprenavir in HIV-1 Infected NNRTI Naive Adults
Brief Title: Investigation of the Potential Pharmacokinetic Interaction Between Nevirapine, Abacavir and Amprenavir in HIV-1 Infected Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) Naive Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1244
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; amprenavir; abacavir

ARMS (3):
- Nevirapine (Experimental): Part I: Study days 15-43
  Part II: Study day 44 to end of trial
  Interventions: Drug: Nevirapine
- Amprenavir (Active Comparator): Part I: Study days 0 to 43
  Part II: Study day 44 to end of trial
  Interventions: Drug: Amprenavir
- Abacavir (Active Comparator): Part I: Study days 0 to 43
  Part II Study day 44 to end of trial
  Interventions: Drug: Abacavir

INTERVENTIONS:
Drug: Nevirapine
  Arms: Nevirapine
Drug: Amprenavir
  Arms: Amprenavir
Drug: Abacavir
  Arms: Abacavir

SUMMARY:
Study to determine the effects of 28 days of nevirapine treatment on the steady-state pharmacokinetics of amprenavir and of abacavir and to further evaluate the pharmacokinetics of nevirapine in combination with amprenavir and abacavir compared to historical controls treated with nevirapine but without amprenavir or abacavir. In addition safety/tolerance of nevirapine, amprenavir and abacavir was to be assessed based on adverse events and clinical laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 65 years, inclusive;
* Plasma HIV-1 RNA >= 5000 copies/mL, documenting HIV-1 infection
* CD4+ cell count >= 100 cells/mm³
* Patients who met the following laboratory parameter:

  * Lymphocyte count >= 1000 cells/mm³
  * Hemoglobin >= 9.0 g/dl (men and women)
  * Platelet count >= 75000 cells/mm3
  * Alkaline Phosphatase <= 3.0 times the upper limit of normal
  * Serum Glutamic-Oxaloacetic Transaminase (SGOT) and Serum Glutamic-Pyruvic Transaminase (SGPT) <= 3.0 times the upper limit of normal
  * Total bilirubin <= 1.5 times the upper limit of normal
  * Creatinine <= 2mg/dL
* Female patients of reproductive potential had to be willing to use a reliable method of double-barrier contraception (such as diaphragm with spermicidal cream or jelly, or condoms with spermicidal foam)
* Patients who were informed of and willing and able to comply with the investigational nature of the study and had signed a written consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Female patients who were pregnant or breast-feeding
* Female patients who intended to change their double-barrier contraception method within 28 days prior to Study Day 0 and throughout the trial
* Patients who in the opinion of the investigator required treatment with a prohibited medication during the study including the potentially toxic substrates such as terfenadine, bepridil, astemizole, cisapride, triazolam, midazolam and ergotamine/dihydroergotamine containing regimes
* Patients taking known inhibitors or inducers of Cytochrome P450 metabolic enzymes including macrolide antibiotics (erythromycin, clarithromycin, azithromycin) azole antifungals (fluconazole, itraconazole) and phenytoin within 28 days prior or Study day 0 and throughout the trial
* Patients receiving immunomodulatory agents
* Ketoconazole, rifabutin and rifampin were excluded during screening and throughout the trial
* Patients with previous exposure to anti-retroviral, such as delavirdine, loviride, efavirenz, nevirapine, abacavir, saquinavir, ritonavir, indinavir, nelfinavir, amprenavir, zidovudine, Lamivudine (3TC), Stavudine (d4T), Didanosine (ddI) and Zalcitabine (ddC)
* Patients receiving any investigational drug or systemic corticosteroids within 30 days of the first dose of study medication and system corticosteroids initially as well as throughout the study and any antineoplastic agent of radiotherapy other than local skin radiotherapy treatment within 12 weeks before starting study medication
* Patients with malabsorption, severe chronic diarrhea or patients unable to maintain adequate oral intake
* Patients currently abusing alcohol or substance abusing; patients on methadone substitution programs might be considered for inclusion in the trial
* Patients undergoing treatment for an active infection
* Patients with hepatic insufficiency due to cirrhosis
* Patients with renal insufficiency
* Patients who were heavy smokers (e.g. > 20 cigarettes per day)
* Patients whose reliability was deemed to put them at risk for non-compliance with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1999-04; Primary Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
AUC (area under plasma concentration time curve) of amprenavir in the absence and presence of nevirapine | Day 14, day 43
Cmax (maximum observed concentration of the analyte in plasma) of amprenavir in the absence and presence of nevirapine | Day 14, day 43
AUC (area under plasma concentration time curve) of abacavir in the absence and presence of nevirapine | Day 14, day 43
Cmax (maximum observed concentration of the analyte in plasma) of abacavir in the absence and presence of nevirapine | Day 14, day 43

SECONDARY OUTCOMES:
Change from baseline in HIV-1 Ribonucleic Acid (RNA) | Baseline, day 14, 21, 28, 35, 43 (Part I), up to 168 days (Part II)
Change from baseline in Lymphocytes Expressing CD4+ cell count | Baseline, day 14, 21, 28, 35, 43 (Part I), up to 168 days (Part II)
Proportion of patients who achieved RNA levels below limit of quantification (BLoQ) (responders) | up to 43 days (Part I), up to 168 days (Part II)
Number of patients with adverse events | up to 240 days
Number of patients with abnormal changes in laboratory parameters | Baseline, day 14, 28, 43 (Part I), up to 168 days (Part II)